CLINICAL TRIAL: NCT01780324
Title: Randomized Clinical Trial of Lidocaine Analgesia for Urethral Catheterization in Children
Brief Title: Lidocaine Analgesia for Urethral Catheterization in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Eileen Klein, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24080004
Record Dates: First submitted 2013-01-17; First posted 2013-01-31 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Pediatric Presentation of Urinary Tract Infection
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No lidocaine (No Intervention): This group will have urinary catheterization without lidocaine (per standard procedure)
- Lidocaine (Experimental): The Intervention is the application of intraurethral lidocaine 5 minutes prior to urethral catheterization.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Intervention - intraurethral lidocaine
  Other Names: lidocaine gel
  Arms: Lidocaine

SUMMARY:
Primary Aim

1. To measure difference in pain via Faces, Legs, Activity, Cry and Consolability (FLACC) Pain Scale score at the time of transurethral bladder catheterization for urine collection in children who do and do not receive intraurethral 2% lidocaine jelly prior to catheterization.

Secondary Aims

1. To assess gender differences in pain control during transurethral bladder catheterization with and without pain control using intraurethral 2% lidocaine jelly.
2. To assess patient discomfort with administration of intraurethral 2% lidocaine jelly.

   To assess parental impression of discomfort between intervention and control groups.
3. To assess pain associated with the administration of intraurethral 2% lidocaine jelly.
4. To measure difference in pain via Modified Behavioral Pain Scale (MBPS) score at the time of TUBC for urine collection in children who do and do not receive intraurethral 2% lidocaine jelly prior to catheterization.

DETAILED DESCRIPTION:
Purpose: To determine whether use of transurethral lidocaine prior to transurethral catheterization for sterile urine collection decreases procedural pain in children 0-3 years old. Primary Aim

1. To measure difference in pain via Faces, Legs, Activity, Cry and Consolability (FLACC) Pain Scale score at the time of transurethral bladder catheterization for urine collection in children who do and do not receive intraurethral 2% lidocaine jelly prior to catheterization.

Secondary Aims

1. To assess gender differences in pain control during transurethral bladder catheterization with and without pain control using intraurethral 2% lidocaine jelly.
2. To assess patient discomfort with administration of intraurethral 2% lidocaine jelly.

   To assess parental impression of discomfort between intervention and control groups.
3. To assess pain associated with the administration of intraurethral 2% lidocaine jelly.
4. To measure difference in pain via Modified Behavioral Pain Scale (MBPS) score at the time of TUBC for urine collection in children who do and do not receive intraurethral 2% lidocaine jelly prior to catheterization.

Rationale: Urinary tract infections (UTIs) are the leading cause of serious bacterial infection in young infants and children. Diagnosis of a UTI in patients in this age group generally requires obtaining a urine sample via transurethral bladder catheterization (TUBC). TUBC is painful, yet standard practice does not include analgesia for infants and children in need of this procedure.

Lidocaine is a commonly used topical anesthetic. Lidocaine jelly can be administered into the urethra prior to catheterization, typically via a preloaded syringe (eg,Uro-Jet) and is FDA approved for this indication. Lidocaine jelly has no antimicrobial characteristics and is a sterile preparation, such that it will not alter urine culture results.

This study is a randomized clinical trial to compare the effectiveness of local 2% lidocaine analgesia instilled in the urethra to reduce the pain and distress in children less than 3 years requiring TUBC.

Reducing the pain and distress associated with TUBC is an important treatment goal, yet there is limited research in children on the effect of intraurethral analgesia during TUBC.

There is growing evidence that children who receive inadequate pain control during invasive procedures may suffer long-term effects.

This Randomized Clinical Trial (RCT) could provide the evidence to drive a change in practice for infants and children requiring bladder catheterization, reducing pain and distress for children undergoing this procedure.

Study Design: This study will enroll 68 children over approximately 1 year. Inclusion criteria includes age 0-3 years, an English or Spanish speaking guardian present to provide consent, and a medical indication for TUBC during the patient's emergency department (ED) visit. Exclusion criteria includes severe developmental delay or impaired mentation; a neural tube defect, paraplegia, or other condition altering urethral sensation; a known urethral stricture, anatomic abnormality or reconstruction; a history of sexual abuse; patient weight less than 2.3 kg; allergy or previous adverse reaction to lidocaine; previous enrollment in the study; or prior successful or attempted TUBC in previous 7 days Subjects will be randomized to receive either usual care for TUBC or 2% lidocaine jelly administered intraurethrally approximately 5 minutes prior to TUBC. Group assignment will be block randomized and stratified by gender. In the lidocaine group, 2% lidocaine would be administered intraurethrally via a blunt tipped Uro-Jet® 5 minutes before TUBC. Lidocaine would not be administered to the usual care group. Both lidocaine administration (if applicable) and TUBC will be videotaped. Research team members will gather information on parental impression of discomfort and patient medical history as well as any adverse events.

A trained, blinded observer will review videotaped procedures and assign pain scores using the Faces, Legs, Activity, Cry and Consolability (FLACC) scale. The FLACC scale is a validated pain scale utilized in pre-verbal children, which assesses pain in 5 separate behaviors during a procedure. For TUBC, pain scores will be recorded at baseline, during catheterization, and one minute after. After assigning FLACC scores, the research team member will then review each video again and assign MBPS scores. MBPS pain scores will be recorded at baseline, during catheterization, and one minute after. Following scoring of the TUBC procedure, patients in the intervention study arm will also have FLACC pain scores assigned one minute before, during, and one minute after administration of lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-3 years
* English or Spanish speaking
* Legal guardian present to provide consent
* Medical indication for TUBC during the patient's ED visit

Exclusion Criteria:

* Severe developmental delay or impaired mentation
* Neural tube defect, paraplegia, or other condition altering urethral sensation
* Known urethral stricture, anatomic abnormality or reconstruction
* History of sexual abuse
* Patient weight less than 2.3 kg
* Allergy or previous adverse reaction to lidocaine
* Previous enrollment in the study
* Prior successful or attempted TUBC in previous 7 days

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Uspal, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 1/30/2013 through 4/27/2014 Location of recruitment: Emergency Department
Pre-assignment Details: All patients consented were randomized.
  186 patients were screened 106 were excluded (41 did not meet inclusion criteria, 52 families declined participation, 13 medical team declined participation, 1 family refused catheterization 80 patients enrolled and randomized
Groups:
- Lidocaine: This group will receive intraurethral lidocaine 5 minutes prior to urethral catheterization.
  Lidocaine gel
Period: Overall Study
Arm/Group | No Lidocaine | Lidocaine
Started | 41 | 39
Completed | 40 | 33
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Lidocaine | Lidocaine | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 39 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 12 (8.1) | 13 (8.5) | 12 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on the Face, Legs, Arms, Cry, Consolability (FLACC) Scale
Description: Pain of urethral catheterization will be determined in the lidocaine and no lidocaine groups. Score range for the FLACC scale was between 0-10 where higher score is more pain.
Time Frame: At time of procedure (up to 30 seconds after catheter insertion)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | No Lidocaine | Lidocaine
Number analyzed (Participants) | 40 | 33
units on a scale | 9 [8 to 10] | 8 [7 to 9]

ADVERSE EVENTS:
Time Frame: Entire study
Arm/Group | No Lidocaine | Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes